CLINICAL TRIAL: NCT01923012
Title: Phase 2 Study Randomized Placebo Controlled With Vitamin K2 in Asymptomatic Calcified Carotid Stenosis
Brief Title: Phase II Randomized Placebo-controlled Study With Vitamin K2 in Asymptomatic Calcified Carotid Stenosis
Acronym: SCAVIT-K2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Sant'Anna (Other)
Responsible Party: Principal Investigator, Simone Vidale, Medical Doctor, Azienda Ospedaliera Sant'Anna
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: OSA-0001
Record Dates: First submitted 2013-08-13; First posted 2013-08-14 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Carotid Disease; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin K2 (Experimental)
  Interventions: Drug: Vitamin K2 (Menaquinone)

INTERVENTIONS:
Drug: Vitamin K2 (Menaquinone)

SUMMARY:
Randomized placebo-controlled study with vitamine K2 (Menaquinone-4) in calcified carotid stenosis. We evaluate the plaque remodelling after administration of vitamine, reducing the calcified component.

ELIGIBILITY:
Inclusion Criteria:

* carotid stenosis between 50 and 70% (NASCET criteria) with calcified plaque

Exclusion Criteria:

* renal and/or hepatic failure
* diseases with secondary calcifications
* dementia
* previous strokes
* concomitant use of anticoagulants
* concomitant infections
* pregnancy or breastfeeding
* reduced patient's compliance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in plaque calcification and carotid stenosis | One year